CLINICAL TRIAL: NCT04679155
Title: Effect of Early vs. Late Eating on Body Composition in Young Adults
Brief Title: Effect of Early Eating on Body Composition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 117951
Record Dates: First submitted 2020-12-16; First posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-11

CONDITIONS: eTRE (Early Time Restricted Eating); lTRE (Late Time Restricted Eating)
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eTRE (Experimental): participants allocated to this group will be required to eat only between 0800h and 1600h.
  Interventions: Behavioral: Eating Time Restriction
- lTRE (Active Comparator): participants allocated to this group will be required to eat only between 1200h and 2000h
  Interventions: Behavioral: Eating Time Restriction

INTERVENTIONS:
Behavioral: Eating Time Restriction — early vs late time of day restriction

SUMMARY:
To our knowledge, as of this day there are only four studies which examined the effects of eTRE with a duration of 12 weeks. There are no studies that examined this phenomenon beyond 12 weeks, one study that lasted five weeks and four studies that lasted 4 weeks or less, some even days. The four studies that lasted 12 weeks in duration all have opportunities to improve upon, which will be discussed here. The first study performed by Gabel et al., focused primarily on measuring body weight, not body composition in older adults. The eating window also began later in the morning at 1000h and finished at 1800h. There also was no restriction on participants consuming caffeine during the fasting window. The second study conducted by Gasmi et al., was focused on strictly older male participants that were active and healthy, again, without measuring body composition. The third study conducted by Wilkinson et al., did not measure body composition and the eating window lasted 10 hours instead of 8. The fourth study performed by Chow et al., examined eTRE with adults aged 45+/-12 years old and did not mention any exclusion criteria based upon physical activity levels or restrictions on caffeine/artificial sweetener intake during the fasting window. Furthermore, none of the studies mentioned above examined eTRE against lTRE directly. We believe that the proposed study will address the concerns mentioned previously and further knowledge associated with eTRE.

DETAILED DESCRIPTION:
Purpose The purpose of the study is to determine the effects of early and late time restricted eating on body composition in overweight and obese young adults. It is hypothesized that early time restricted eating will provide a more desirable effect (lower fat mass) on body composition for the participants.

Sample The sample will include 30 overweight/obese young adults, male and female, ranging in age from 18-30 that volunteer to participate in the study. This sample size is justified assuming a standard deviation of 1.5 based on previous studies and using a power of 80% with the statistical significance of 0.05 the resulting n would be 2(1.5)^2*(0.84+1.96)^2/5=7 (Kadam, P., & Bhalerao, S. (2010). Sample size calculation. International journal of Ayurveda research, 1(1), 55). To account for dropouts/non-interest in participation, 10 participants will be recruited for each group. All individuals must give written informed consent in order to participate in the study. Exclusion criteria include self-reported: diabetes, smoking, CVD, pregnancy, weight loss medication, physical activity level greater than low/sedentary (7500 steps daily), unstable weight (>4kg loss/gain) for 3 months prior to study commencement.

Procedure Inclusion/exclusion criteria will be explicitly stated throughout the recruitment process. Potential participants will be recruited through mass email recruitment via Western email services, presenting one-slide information sessions at the beginning of lectures and posting flyers around campus. Participants will then be in direct contact with Reed Zehr to set up a meeting to gain information of the study. After the information meeting the individuals will be given up to 3 days to determine if they want to participate and give their informed consent. See attached form in the consent section of the ethics application.

Measurement: All participants will be required to have their Body Composition measured using non-invasive densitometry (BodPod). The procedure poses no risk to the participant and takes approximately 5 minutes to complete. This procedure will take place initially one week prior to study commencement and then every 4 weeks after study commencement until the 12 weeks of the study duration are complete. This results in a total of 4 measurements. Upper body strength measurements will be recorded one week prior to commencement of the study and once again after study completion using a maximal bench press test. Lower body strength measurements will be recorded one week prior to commencement of the study and once again after study completion using a maximal leg press test. Completion of a health-related quality of life questionnaire one week prior to commencement of the study and once again after study completion is also required.

ELIGIBILITY:
Inclusion Criteria:

* sedentary- lightly physically active (<7,500 steps daily)
* BMI > 25
* 18-30 yo.

Exclusion Criteria:

* Have diabetes (self-reported)
* Have history of smoking (self-reported)
* Have history of cardiovascular disease (self-reported)
* Have BMI of <24.9
* Are pregnant or become pregnant during the study (self-reported)
* Take medication for weight loss (self-reported)
* Physical activity level > 7500 steps/day
* Unstable weight for 3 months prior to commencement of study (>4kg weight loss/gain)
* Employed in a shift work position

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Body Composition | <5 mins
  fat mass vs. fat-free mass via BodPod

SECONDARY OUTCOMES:
upper body strength test | <10 mins
  1 rep maximal progressive loading bench press test
lower body strength test | <10 mins
  1 rep maximal progressive loading leg press test
health related quality of life questionnaire | <10 mins
  subjective feelings of overall health per participant

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Nutrition Laboratory, Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No